CLINICAL TRIAL: NCT02397161
Title: Improving Mental Attention, Timing of Muscle Activation and Reactive Balance Control in Children With Developmental Coordination Disorder: A Randomized Controlled Trial
Brief Title: Mental Attention-neuromuscular Training for Children With Developmental Coordination Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shirley S.M. Fong, Assistant Professor, DRPC chairperson, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17120515
Record Dates: First submitted 2015-03-09; First posted 2015-03-24 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Developmental Coordination Disorder
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- AT-NMT (Experimental): AT-NMT group - will receive a 12-week EEG biofeedback mental attention-neuromuscular training
  Interventions: Other: EEG biofeedback mental attention-neuromuscular training
- NMT alone (Experimental): NMT group - will receive a 12-week neuromuscular training
  Interventions: Other: Neuromuscular training
- AT alone (Experimental): AT group - will receive a 12-week EEG biofeedback mental attention training
  Interventions: Other: EEG biofeedback mental attention training
- Control (No Intervention): Control group - no intervention for 12 weeks

INTERVENTIONS:
Other: EEG biofeedback mental attention-neuromuscular training — Mental attention training using EEG biofeedback and neuromuscular training using physio-therapeutic exercises
  Arms: AT-NMT
Other: Neuromuscular training — Neuromuscular training using physio-therapeutic exercises
  Arms: NMT alone
Other: EEG biofeedback mental attention training — Mental attention training using EEG biofeedback
  Arms: AT alone

SUMMARY:
Objective: To compare the effectiveness of EEG biofeedback mental attention-neuromuscular training (AT-NMT), neuromuscular training (NMT) alone, EEG biofeedback mental attention training (AT) alone, and no intervention for improving reactive balance performance among children with developmental coordination disorder (DCD).

Design: A single-blinded, randomized controlled clinical trial. Sample: 172 children with DCD. Interventions: AT-NMT, NMT, AT, or no intervention for 12 weeks. Major outcomes: Outcomes will be evaluated at baseline, post-intervention, and 3-month follow-up. A motor control test (MCT) will give a composite latency score, prefrontal cortex EEG recordings during MCT will measure the mental attention level, and surface electromyography recordings during MCT will indicate the lower limb muscle onset latency.

DETAILED DESCRIPTION:
Hypothesis: The Investigators hypothesize that the reactive balance performance in children with DCD can be best improved by treating both their mental attention and neuromuscular deficits.

Objective: To compare the effectiveness of AT-NMT, NMT alone, AT alone, and no intervention for improving reactive balance performance among children with DCD.

Design: A single-blinded, randomized controlled clinical trial. Sample: 172 children with DCD. Interventions: AT-NMT, NMT, AT, or no intervention for 12 weeks. Major outcomes: Outcomes will be evaluated at baseline, post-intervention, and 3-month follow-up. A motor control test (MCT) will give a composite latency score, prefrontal cortex EEG recordings during MCT will measure the mental attention level, and surface electromyography recordings during MCT will indicate the lower limb muscle onset latency.

Anticipated results and clinical significance: Children with DCD who receive AT-NMT will have the best reactive balance performance outcomes. If the results are positive, this novel training regime can be readily adopted in clinical practice. AT-NMT will improve overall well-being in these children and have positive socio-economic implications such as shorter rehabilitation periods and reduced healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

1. 6 to 9 years old;
2. a formal diagnosis of DCD based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) at a child assessment center;
3. a Bruininks-Oseretsky Test of Motor Proficiency giving a gross motor composite score of ≤42;
4. a Child Behavior Checklist attention problem subscale T score of ≥54.5, indicating an attention deficit;
5. attending a local mainstream school;
6. an intelligence level within the normal range; and
7. no experience in using the Brain Computer Interface system or similar apparatus.

Exclusion Criteria:

1. a diagnosis of neurological or other movement disorder;
2. any cognitive, psychiatric (comorbid ADHD will not be excluded), congenital, musculoskeletal or cardiopulmonary disorder that can affect motor performance;
3. receiving active therapies or treatments including complementary and alternative medicine;
4. demonstrating excessive disruptive behavior; or
5. those unable to follow instructions adequately.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change in motor control test composite latency score | Baseline (0 month), post-intervention (3 months), and 3-month follow-up (6 months)

SECONDARY OUTCOMES:
Change in EEG mental attention level | Baseline (0 month), post-intervention (3 months), and 3-month follow-up (6 months)
Change in surface EMG lower limb muscle onset latency | Baseline (0 month), post-intervention (3 months), and 3-month follow-up (6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley SM Fong, PT, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Pokfulam, Hong Kong